CLINICAL TRIAL: NCT05184751
Title: Incidence and Risk Factors of Early Onset Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Hospital Frydek-Mistek (Other)
Responsible Party: Principal Investigator, Ivana Mikoviny Kajzrlikova, MD, PhD, MD, PhD, Head of endoscopic department, Hospital Frydek-Mistek
Other Study IDs: Early onset colorectal cancer
Record Dates: First submitted 2021-12-22; First posted 2022-01-11 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 50 years and over: patients who underwent colonoscopic examination aged 50 years and over
  Interventions: Other: colonoscopy
- under 50 years: patients who underwent colonoscopic examination aged under 50 years
  Interventions: Other: colonoscopy

INTERVENTIONS:
Other: colonoscopy

SUMMARY:
Early onset colorectal cancer (cancer in person younger than 50 years) has increasing incidence last years. The aim of our study was to assess the real-life incidence of early onset colorectal cancer, advanced neoplasias (colorectal cancer and/or advanced adenoma) and all neoplastic lesions in total in a single non-university endoscopic center.

DETAILED DESCRIPTION:
The investigators retrospectively assessed the incidence of all neoplastic lesions, advanced neoplasias and colorectal cancer in population under 50 years of age compared to population 50 years and older. The investigators collected the data from all colonoscopic examinations performed in non-university hospital Frydek-Mistek from January 2012 to the end of June 2021.

ELIGIBILITY:
Inclusion Criteria: all patient who underwent colonoscopic examination clear indication for colonoscopy

Exclusion Criteria: not able to underwent colonoscopy

Ages: 4 Years to 97 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: all patients who were indicated for colonoscopic examination (all indications) in period january 2012 to the end of june 2021
Sampling Method: Probability Sample
Enrollment: 18257 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
incidence of early onset colorectal neoplasias, risk factors | 10 years
  the real-life incidence of early onset colorectal cancer, advanced neoplasias (colorectal cancer and/or advanced adenoma) and all neoplastic lesions in total in a single non-university endoscopic center, the risk of sex and family history of colorectal cancer

CONTACTS AND LOCATIONS:
Overall Officials: Ivana Mikoviny Kajzrlikova, Principal Investigator — Hospital Frydek-Mistek

IPD SHARING:
Plan to Share IPD: Undecided